CLINICAL TRIAL: NCT06590532
Title: French Randomised Controlled Trial Investigating the Clinical and Cost-effectiveness Role of a Cloud-based, Artificial Intelligent Image Fusion System to Guide Endovascular Aortic Aneurysm Repair and Aorto Iliac Revascularisation.
Brief Title: Evaluation of the Clinical and Cost-effectiveness of an Automated Mobile Hybrid Room in Vascular Surgery Compared with Current Practice
Acronym: RADIOPROTEC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC22_0396
Record Dates: First submitted 2024-06-24; First posted 2024-09-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Endovascular
MeSH Terms: interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fusion group (Experimental): patient undergoing endovascular aortic repair with fusion imaging system guidance
  Interventions: Procedure: Endovascular aneurysm repair or aorto iliac endovascular revascularisation with Fusion imaging system Cydar-EV
- Control group (Active Comparator): patient undergoing endovascular aortic repair without fusion imaging system guidance (only with X-rays and roadmaping)
  Interventions: Procedure: Endovascular aneurysm repair or aorto iliac endovascular revascularisation without Fusion imaging system Cydar-EV

INTERVENTIONS:
Procedure: Endovascular aneurysm repair or aorto iliac endovascular revascularisation with Fusion imaging system Cydar-EV — Cydar-EV image fusion is a CE-marked medical device, which instead of a table-tacked overlay uses computer vision to fuse pre-procedural 3D images with intra-operative 2D fluoroscopy automatically and in real-time.
  Arms: Fusion group
Procedure: Endovascular aneurysm repair or aorto iliac endovascular revascularisation without Fusion imaging system Cydar-EV — patients will be assigned either to an endovascular repair using standard X-ray fluoroscopy imaging alone (the current reference standard)
  Arms: Control group

SUMMARY:
Evaluation of the clinical and cost-effectiveness of a mobile hybrid room compared with current practice without mobile hybrid room and imaging fusion guidance, in a French multicentre clinical setting.

The hypothesis is that the use of a mobile hybrid room with an automated artificial intelligent image fusion system would directly benefit patients, health worker and health care system by reducing procedure time, patient and staff exposure to radiation, improve clinical success and reduce costs (requested by a fixed imaging system installation and increasing the number of patients). This will also improve the safety of these procedures for patient and staff, when a conventional hybrid room is not available

DETAILED DESCRIPTION:
Multi-centre, patient- and observer-blinded, two-armed, parallel groups randomised controlled trial. 7 French University hospital will include 350 patients presenting with AAA or aorto iliac occlusive disease suitable for endovascular treatment, to either repair using standard X-ray fluoroscopy imaging alone (the current reference standard) or augmented with automated image fusion. The study will be conducted in real-world clinical settings and will focus on multiple providers to demonstrate the effect in the wider healthcare system.

The trial will be conducted in 7 centres in France over 24 months. 350 patients will be recruited over a 18 month period, with 3 months minimum follow-up. Every vascular surgeon will be trained to use properly the fusion system, and the first 5 patients of each center won't be included.

Radiation parameters (machine report, passive dosimeters), iodinated contrast, technical and clinical success at 30-d and 3 months, procedure time, fluoro time, and costs will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Procedure carried out in an operating theatre equipped with a mobile operating theatre C-arm or a mobile planar or an old-generation fixed room with no image fusion available
* Surgeon trained in the use of image fusion
* Operator who has given their consent
* Endovascular management of an aorto-iliac artery disease or a sub-renal AAA using a sub-renal bifurcated stent graft
* Patient in possession of an angioscan less than 6 months old
* Patient of legal age who has given his/her consent
* Ionising radiation generator with up-to-date and validated quality control
* Participant affiliated to a Social Security scheme

Exclusion Criteria:

* First procedure with fusion for the previously trained surgeon.
* Procedure performed without an operating aid.
* Emergency procedure.
* Associated surgical procedure (femoropopliteal lesions, lesions of the renal or digestive arteries, iliac branch).

digestive arteries, iliac branch).

* Patients with AAA that cannot be treated by a simple sub-renal endovascular approach simple endovascular approach (subrenal bifurcated stent graft)
* Aortic emergencies (ruptured AAA).
* Persons under guardianship, curatorship or safeguard of justice
* Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Cost consequence analysis associated with endovascular procedures performed using automatic imaging fusion guidance and conventional endovascular technique performed without image fusion guidance up to 30 days time horizon and a collective perspective. | 18 month
  To compare the costs and consequences associated with endovascular procedures performed using automatic imaging fusion guidance and conventional endovascular technique performed without image fusion guidance. Consequences are listed in the secondary endpoints. Cos twill be express in €.

SECONDARY OUTCOMES:
X-ray dose per procedure | day 0
  exposure parameters from the machine
X-ray dose per procedure for the physician | day 0
  exposure parameters from the dosimeter
Contrast dose per procedure | day 0
  Contrast dose used
Length of ITU/HDU admission | 18 months
  Length of ITU/HDU admission
Technical success | day 0
  defined as proximal and distal seal zone at least 10mm and no evidence of endoleak or revascularization success.
Clinical success | 1 month
  defined as primary patency rate or endovascular exclusion of the aneurysm
30-day mortality | 30 days
  30-day mortality
Quality of life questionnaire | 30 days
  EQ-5D-5L assessement
cost-effectiveness | 5 years
  Net financial impact over 5 years of SHMA deployment (based on the 5-year projection and different different scenarios for the spread of the technology)

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Rinckenbach, Besançon, Besançon
  - NASR, Brest, Brest
  - El Batti, Créteil, Créteil
  - Spear, Grenoble, Grenoble
  - Pr Blandine Maurel, Nantes, Nantes
  - Jean-Baptiste, Nice, Nice
  - Duprey, Reims, Reims

IPD SHARING:
Plan to Share IPD: No